CLINICAL TRIAL: NCT00252720
Title: DIRECT: DIabetic Retinopathy Candesartan Trials. Effects of Candesartan Cilexetil (Candesartan) on Diabetic Retinopathy in Type 1 Diabetic Patients With Retinopathy.
Brief Title: DIabetic Retinopathy Candesartan Trials.
Acronym: DIRECT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D2453C00046; DIRECT; SH-AHM-0046
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Results first posted 2014-06-03 (Estimated); Last update posted 2014-06-03 (Estimated); Status verified 2014-04

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes mellitus type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — candesartan; candesartan cilexetil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- candesartan (Experimental): candesartan cilexetil 32 mg once daily
  Interventions: Drug: candesartan
- placebo (No Intervention): control

INTERVENTIONS:
Drug: candesartan — 32 mg oral tablet
  Other Names: ATACAND
  Arms: candesartan

SUMMARY:
The primary objective is to determine whether candesartan, compared to placebo reduces the progression of diabetic retinopathy in normotensive, normoalbuminuric type 1 diabetic patients with retinopathy.

The secondary objective is to determine whether candesartan, compared to placebo, reduces the incidence of clinically significant macular oedema (CSME) and/or proliferative diabetic retinopathy (PDR) and beneficially influences the rate of change in urinary albumin excretion rate (UAER).

This study is part of the DIRECT Programme also including a primary prevention study of diabetic retinopathy in type 1 diabetes and a secondary prevention study in type 2 diabetes. The primary objective for all three pooled studies is to determine whether candesartan, compared to placebo, reduces the incidence of microalbuminuria in type 1 and type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18 - 55 years with type 1 diabetes diagnosed before age of 36 years and in need for continuous insulin treatment within 1 year of diagnosis of diabetes are included.
* Duration of diabetes for > 1 year and < 20 years with stable diabetic therapy within last 6 months.
* Patients with untreated resting mean sitting SBP < 130 mmHg, mean sitting DBP < 85 mmHg and with retinal photograph grading level > 20/10 up to < 47/47 (on ETDRS severity scale).

Exclusion Criteria:

* Patients with the following conditions are excluded from participation on the study:
* Cataract or media opacity of a degree which precludes taking gradable retinal photographs
* Angle closure glaucoma, which precludes pharmacological dilatation of the pupil
* History or presence of proliferative retinopathy
* History or presence of clinical significant macular oedema (CSME)
* History or evidence of photocoagulation of the retina
* Other retinal conditions which may mask assessment, eg, retinal vein occlusion
* Positive micral dipstick test
* Presence of secondary diabetes
* Pregnant or lactating women or women of child bearing potential not practicing an adequate method of contraception
* Need of treatment with ACE-inhibitor
* Haemodynamically significant aortic or mitral valve stenosis
* Known renal artery stenosis or kidney transplantation
* Hypersensitivity to study drug
* Severe concomitant disease which may interfere with the assessment of the patient, eg, malignancy, as judged by the investigator

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1850 (Actual)
Dates: Start 2001-08; Primary Completion 2008-02 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Atacand Medical Science Director, MD, Study Director — AstraZeneca

REFERENCES:
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] Sjolie AK, Klein R, Porta M, Orchard T, Fuller J, Parving HH, Bilous R, Aldington S, Chaturvedi N. Retinal microaneurysm count predicts progression and regression of diabetic retinopathy. Post-hoc results from the DIRECT Programme. Diabet Med. 2011 Mar;28(3):345-51. doi: 10.1111/j.1464-5491.2010.03210.x. PMID 21309844
- [Derived] Porta M, Hainer JW, Jansson SO, Malm A, Bilous R, Chaturvedi N, Fuller JH, Klein R, Orchard T, Parving HH, Sjolie AK; DIRECT Study Group. Exposure to candesartan during the first trimester of pregnancy in type 1 diabetes: experience from the placebo-controlled DIabetic REtinopathy Candesartan Trials. Diabetologia. 2011 Jun;54(6):1298-303. doi: 10.1007/s00125-010-2040-1. Epub 2011 Jan 12. PMID 21225239
- [Derived] Bilous R, Chaturvedi N, Sjolie AK, Fuller J, Klein R, Orchard T, Porta M, Parving HH. Effect of candesartan on microalbuminuria and albumin excretion rate in diabetes: three randomized trials. Ann Intern Med. 2009 Jul 7;151(1):11-20, W3-4. doi: 10.7326/0003-4819-151-1-200907070-00120. Epub 2009 May 18. PMID 19451554
- [Derived] Chaturvedi N, Porta M, Klein R, Orchard T, Fuller J, Parving HH, Bilous R, Sjolie AK; DIRECT Programme Study Group. Effect of candesartan on prevention (DIRECT-Prevent 1) and progression (DIRECT-Protect 1) of retinopathy in type 1 diabetes: randomised, placebo-controlled trials. Lancet. 2008 Oct 18;372(9647):1394-402. doi: 10.1016/S0140-6736(08)61412-9. Epub 2008 Sep 25. PMID 18823656
- See also: Related Info — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1268&filename=CSR-D2453C00046.pdf
- See also: CSR-D2453C00046.pdf — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_6111&studyid=1268&filename=CSR-D2453C00046.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled in the DIRECT programme 8 June 2001 and last subject completed the DIRECT programme 16 April 2008 mainly in hospital based clinics. The study investigators enrolled 4514 patients with type 1 diabetes to either Study 45 or 46, of whom 1905 proceeded to randomization into Study 46 (1421 into Study 45).
Pre-assignment Details: The most common reason for not being randomized was that all eligibility criteria were not fulfilled, followed by withdrawn informed consent.
Groups:
- Placebo: Placebo Comparator
Period: Overall Study
Arm/Group | Candesartan | Placebo
Started | 951 | 954
Completed | 819 | 789
Not Completed | 132 | 165
Not completed — Withdrawal by Subject | 95 | 97
Not completed — Death | 7 | 8
Not completed — Moving | 23 | 42
Not completed — Mainly patients lost to follow-up | 7 | 18

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Candesartan | Placebo | Total
Number analyzed (Participants) | 951 | 954 | 1905
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 951 | 954 | 1905
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (8.5) | 31.9 (8.5) | 31.7 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 413 | 401 | 814
  Male | 538 | 553 | 1091
Region of Enrollment [Number; unit: participants]
  Russian Federation | 186 | 162 | 348
  Europe | 595 | 619 | 1214
  Canada | 69 | 71 | 140
  South Africa | 101 | 102 | 203

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a 3-step or Greater Increase in Early Treatment of Diabetic Retinopathy Study (EDTRS) Severity Scale
Description: Retinopathy progression was defined as the first occurrence of at least a 3-step increase in the ETDRS severity scale. 3 steps were defined as either a 1-step change in one eye and a 2-step change in the other eye or as a 3-step change in one eye only. EDRTS is a scale with 11 steps (1-11). A generlized log-rank test was used to test difference between treatments.
Time Frame: From baseline to end of study, i.e. 5 years, with visits after a half year, one year and thereafter one visit per year.
Population: The population was the Intention to Treat population which includes all randomized patients with any post-randomization data.
Measure: Number; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
Participants | 127 (0.034) | 124 (0.033)
Statistical Analysis 1: Comparison: Candesartan vs Placebo; Test type: Superiority or Other; p = 0.8487, Log Rank; Generalized; Hazard Ratio (HR) = 1.024, 95% CI 2-sided [0.800 to 1.312]

2. Secondary Outcome: Number of Participants With a Regression of Diabetic Retinopathy.
Description: Regression of diabetic retinopathy was defined as at least a 3 step improvement or a persistent 2-step improvement (confirmed in 2 consecutive photography sets) in the Early Treatment of Diabetic Retinopathy Study (ETDRS) severity scale. 3 steps were defined as either a 1-step change in one eye and a 2-step change in the other eye or as a 3-step change in one eye only. EDRTS is a scale with 11 steps (1-11).
Time Frame: From baseline to the end of the study, i.e., 5 years
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
Participants | 140 (0.039) | 139 (0.039)

3. Secondary Outcome: Number of Participants With Incident Clinically Significant Macular Edema (CSME) and/or Proliferative Diabetic Retinopathy (PDR).
Description: Clinically Significant Macular Edema (CSME) and Proliferative Diabetic Retinopathy (PDR) are diagnosed via retinal photographs.
Time Frame: From baseline to end of study, i.e. 5 years.
Population: The population was the Intention To Treat population whick includes all randomized patients with any post-randomization data.
Measure: Number; unit: Participants
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
Participants | 110 (0.03) | 107 (0.03)

4. Secondary Outcome: Rate of Change in Urinary Albumin Excretion Rate (UAER).
Description: An estimate of the slope from fitting a linear regression of log (UAER) over time (post-randimisation, yearly assessments) for each patient
Time Frame: From baseline to end of study, i.e. 5 years.
Population: The population was the Intention To Treat population which includes all randimized patients with any post-randomization data.
Measure: Least Squares Mean (95% Confidence Interval); unit: log (µg/min)/year
Arm/Group | Candesartan | Placebo
Number analyzed (Participants) | 951 | 954
log (µg/min)/year | 0.569 [0.489 to 0.648] | 0.642 [0.563 to 0.722]

ADVERSE EVENTS:
Time Frame: During treatment. During Treatment refers to the period of actual treatment with randomized study drug, ie, is a subset of the patients included in During Study. During Treatment period only includes AEs reported while patients were on study treatment.
Description: Population used was the safety population which includes all patients who received at least 1 dose of randomized study strug and for whom any post-dose data were available.
Arm/Group | Candesartan | Placebo
Serious Adverse Events (participants affected / at risk) | 173/951 | 161/951
Other Adverse Events (participants affected / at risk) | 92/951 | 32/951
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan (N=951) | Placebo (N=951)
Idiopathic Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 1
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenic Purpura (Blood and lymphatic system disorders) | 1 | 0
Myocardial Infarction (Cardiac disorders) | 1 | 2
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Angina Pectoris (Cardiac disorders) | 0 | 1
Cardiovascular Disorder (Cardiac disorders) | 0 | 1
Heart Disease Congenital (Congenital, familial and genetic disorders) | 0 | 1
Hepato-Lenticular Degeneration (Congenital, familial and genetic disorders) | 0 | 1
Ear Congestion (Ear and labyrinth disorders) | 0 | 1
Sudden Hearing Loss (Ear and labyrinth disorders) | 0 | 1
Vestibular Neuronitis (Ear and labyrinth disorders) | 1 | 0
Addison's Disease (Endocrine disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 1 | 0
Diabetic Blindness (Eye disorders) | 0 | 1
Eye Haemorrhage (Eye disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 5 | 2
Abdominal Pain (Gastrointestinal disorders) | 2 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 2
Abdominal Adhesions (Gastrointestinal disorders) | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Anal Fissure (Gastrointestinal disorders) | 1 | 0
Change Of Bowel Habit (Gastrointestinal disorders) | 0 | 1
Coeliac Disease (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Duodenal Ulcer Perforation (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 1
Food Poisoning (Gastrointestinal disorders) | 0 | 1
Gastric Ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1
Gingival Disorder (Gastrointestinal disorders) | 0 | 1
Hiatus Hernia (Gastrointestinal disorders) | 0 | 1
Irritable Bowel Syndrome (Gastrointestinal disorders) | 1 | 0
Pancreatitis Acute (Gastrointestinal disorders) | 0 | 1
Rectal Polyp (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0
Chest Pain (General disorders) | 5 | 0
Death (General disorders) | 0 | 1
Foreign Body Reaction (General disorders) | 0 | 1
Macrosomia (General disorders) | 0 | 1
Oedema (General disorders) | 1 | 0
Oedema Peripheral (General disorders) | 1 | 0
Organ Failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 1
Hepatitis Acute (Hepatobiliary disorders) | 0 | 1
Hepatitis Toxic (Hepatobiliary disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
Appendicitis (Infections and infestations) | 4 | 4
Gastroenteritis (Infections and infestations) | 2 | 3
Pneumonia (Infections and infestations) | 3 | 3
Pyelonephritis Acute (Infections and infestations) | 3 | 1
Respiratory Tract Infection (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 1 | 2
Hepatitis B (Infections and infestations) | 2 | 0
Localised Infection (Infections and infestations) | 2 | 0
Pilonidal Cyst (Infections and infestations) | 2 | 0
Postoperative Wound Infection (Infections and infestations) | 2 | 0
Pyelonephritis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 2 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 2 | 1
Viral Infection (Infections and infestations) | 1 | 2
Abdominal Abscess (Infections and infestations) | 0 | 1
Abdominal Wall Abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess Limb (Infections and infestations) | 0 | 1
Acute Tonsillitis (Infections and infestations) | 0 | 1
Adnexitis (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Corneal Infection (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 1 | 0
Encephalitis Viral (Infections and infestations) | 0 | 1
Gastrointestinal Infection (Infections and infestations) | 0 | 1
Groin Abscess (Infections and infestations) | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0
Hepatitis C (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 0 | 1
Infected Cyst (Infections and infestations) | 1 | 0
Liver Abscess (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 1 | 1
Oophoritis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Pelvic Inflammatory Disease (Infections and infestations) | 0 | 1
Perianal Abscess (Infections and infestations) | 1 | 1
Perineal Abscess (Infections and infestations) | 1 | 0
Peritonsillar Abscess (Infections and infestations) | 1 | 1
Pulmonary Tuberculosis (Infections and infestations) | 1 | 0
Pyelonephritis Chronic (Infections and infestations) | 0 | 1
Retroperitoneal Abscess (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Viral Diarrhoea (Infections and infestations) | 1 | 0
Viral Skin Infection (Infections and infestations) | 0 | 1
Wound Infection Staphylococcal (Infections and infestations) | 1 | 0
Road Traffic Accident (Injury, poisoning and procedural complications) | 4 | 2
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 3
Multiple Injuries (Injury, poisoning and procedural complications) | 2 | 3
Hand Fracture (Injury, poisoning and procedural complications) | 2 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 2 | 0
Ligament Injury (Injury, poisoning and procedural complications) | 0 | 2
Lower Limb Fracture (Injury, poisoning and procedural complications) | 2 | 2
Overdose (Injury, poisoning and procedural complications) | 1 | 2
Accidental Overdose (Injury, poisoning and procedural complications) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 1 | 0
Cartilage Injury (Injury, poisoning and procedural complications) | 1 | 1
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Epicondylitis (Injury, poisoning and procedural complications) | 0 | 1
Femur Fracture (Injury, poisoning and procedural complications) | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 1 | 0
Frostbite (Injury, poisoning and procedural complications) | 0 | 1
Gun Shot Wound (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 1 | 0
Injury Corneal (Injury, poisoning and procedural complications) | 0 | 1
Intentional Overdose (Injury, poisoning and procedural complications) | 1 | 0
Intervertebral Disc Injury (Injury, poisoning and procedural complications) | 1 | 0
Joint Dislocation (Injury, poisoning and procedural complications) | 1 | 0
Joint Injury (Injury, poisoning and procedural complications) | 0 | 1
Ligament Rupture (Injury, poisoning and procedural complications) | 1 | 0
Limb Injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple Fractures (Injury, poisoning and procedural complications) | 0 | 1
Patella Fracture (Injury, poisoning and procedural complications) | 0 | 1
Radius Fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 0 | 1
Skull Fractured Base (Injury, poisoning and procedural complications) | 1 | 0
Sports Injury (Injury, poisoning and procedural complications) | 1 | 0
Tendon Injury (Injury, poisoning and procedural complications) | 1 | 0
Thermal Burn (Injury, poisoning and procedural complications) | 0 | 1
Tibia Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hepatitis C Positive (Investigations) | 0 | 1
Tumour Marker Increased (Investigations) | 0 | 1
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 26 | 17
Hypoglycaemia (Metabolism and nutrition disorders) | 16 | 24
Hyperglycaemia (Metabolism and nutrition disorders) | 8 | 13
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 11 | 8
Ketoacidosis (Metabolism and nutrition disorders) | 1 | 6
Hypoglycaemic Seizure (Metabolism and nutrition disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Diabetic Foot (Metabolism and nutrition disorders) | 1 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dupuytren's Contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Trigger Finger (Musculoskeletal and connective tissue disorders) | 1 | 1
Fibroadenoma Of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Malignant Melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Anaplastic Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign Colonic Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary Thyroid Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Penile Wart (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypoglycaemic Coma (Nervous system disorders) | 3 | 5
Carpal Tunnel Syndrome (Nervous system disorders) | 4 | 1
Diabetic Coma (Nervous system disorders) | 2 | 0
Diabetic Neuropathy (Nervous system disorders) | 0 | 2
Grand Mal Convulsion (Nervous system disorders) | 2 | 1
Amnesia (Nervous system disorders) | 1 | 0
Cerebral Haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular Accident (Nervous system disorders) | 1 | 1
Diabetic Hyperosmolar Coma (Nervous system disorders) | 1 | 0
Diabetic Ketoacidotic Hyperglycaemic Coma (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 1 | 0
Haemorrhagic Stroke (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Multiple Sclerosis (Nervous system disorders) | 1 | 0
Myelitis (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Tension Headache (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Foetal Cardiac Disorder (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Intra-Uterine Death (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Major Depression (Psychiatric disorders) | 0 | 1
Suicide Attempt (Psychiatric disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 2 | 0
Calculus Urinary (Renal and urinary disorders) | 1 | 0
Diabetic Nephropathy (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal Failure (Renal and urinary disorders) | 0 | 1
Ureteric Stenosis (Renal and urinary disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 2
Cervical Dysplasia (Reproductive system and breast disorders) | 1 | 0
Dysfunctional Uterine Bleeding (Reproductive system and breast disorders) | 0 | 1
Endometriosis (Reproductive system and breast disorders) | 1 | 0
Menometrorrhagia (Reproductive system and breast disorders) | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 1 | 1
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 1
Pelvic Pain (Reproductive system and breast disorders) | 0 | 1
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 1 | 0
Bronchitis Chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Polyps (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal Septum Deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal Cord Polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema Nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Skin Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Femoral Artery Occlusion (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 0 | 1
Varicose Vein (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Candesartan (N=951) | Placebo (N=951)
Hypotension (Vascular disorders) | 92 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No